CLINICAL TRIAL: NCT00422019
Title: A Global, Multicenter, Open-label, Single Agent, Two-stage Phase 2 Study to Evaluate the Efficacy and Safety of AMG 102 in Subjects With Advanced Renal Cell Carcinoma
Brief Title: A Phase II Study to Treat Subjects With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060100
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: Renal Cancer; Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

ARMS (2):
- AMG 102 at 20 mg/kg Dose Level (Experimental): Up to 40 subjects will be treated at 20 mg/kg of AMG 102 Q2W (every 2 weeks) depending upon the stage of the study and number of responses observed.
  Interventions: Drug: AMG 102 at 20 mg/kg
- AMG 102 at 10 mg/kg Dose Level (Experimental): Up to 40 subjects will be dosed at 10mg/kg of AMG 102 Q2W (every two weeks) based upon the stage of the study and number of responses observed.
  Interventions: Drug: AMG 102 at 10 mg/kg

INTERVENTIONS:
Drug: AMG 102 at 10 mg/kg — AMG 102 at 10 mg/kg IV (in the vein) every 2 weeks
  Arms: AMG 102 at 10 mg/kg Dose Level
Drug: AMG 102 at 20 mg/kg — AMG 102 at 20 mg/kg IV (in the vein) every 2 weeks
  Arms: AMG 102 at 20 mg/kg Dose Level

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of AMG 102 in patients with Advanced Renal Cancer.

ELIGIBILITY:
Inclusion Criteria:

* documented histologically confirmed advanced or metastatic renal cell carcinoma with the primary tumor in place or following nephrectomy
* measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques (CT or MRI) or ≥ 10 mm by spiral CT scan
* no more than 3 relapses (or prior systemic treatments)
* unable to receive or failed prior therapy with vascular endothelial growth factor (VEGF) binding agents or VEGF receptor tyrosine kinase inhibitors or other multi-kinase inhibitors
* tissue blocks or tissue sections from initial or upon diagnosis of advanced metastatic disease are available for submission to the central laboratory within approximately 4 weeks after enrollment or approval is granted by the sponsor (upon receipt of justification why the sample is not available)
* age ≥ 18 years
* ECOG performance status of 0-2
* hemoglobin concentration ≥ 9 g/dL
* absolute neutrophil count ≥ 1.5 x 10(9th)/L
* corrected serum calcium ≤ 10 mg/dL
* either serum creatinine < 2.0 x upper limit of normal OR creatinine clearance > 40 mL/min
* alanine aminotransferase ≤ 2.5 times upper limit of normal or < 5.0 x ULN if the subject has documented liver metastasis or primary hepatic neoplasm
* serum total bilirubin ≤ 2.5 times upper limit of normal
* before any study-specific procedure, the appropriate written informed consent must be obtained

Exclusion Criteria:

* active brain metastases; brain metastases allowed provided they have been treated with surgery and/or radiation therapy and show no evidence of progression on cerebral CT or MRI scan 2 months following surgery and/or radiation therapy
* concurrent severe and/or uncontrolled medical disease (e.g., uncontrolled diabetes, congestive cardiac failure, myocardial infarction within 6 months before enrollment) that could compromise participation in the study
* documented history of human immunodeficiency virus infection
* documented history of viral chronic hepatitis
* received biologic, small molecule, immunotherapy, chemotherapy, radiotherapy or other agents to treat renal cancer within 28 days before enrollment
* treated previously with c-Met or HGF targeted therapy
* concurrent or prior (within 7 days before enrollment) anticoagulation therapy, except:

  * Use of low-dose warfarin (< 2 mg/day) for prophylaxis against central venous catheter thrombosis or
  * Use of low molecular weight heparins (LMWH, e.g., enoxaparin sodium [Lovenox] and unfractionated heparin for prophylaxis against central venous catheter thrombosis is allowed
* concurrent use of hormones or other chemotherapeutic agents except for steroids given for adrenal failure and hormones administered for non-disease-related conditions (eg, insulin for diabetes); except for non-cancer reasons
* concurrent palliative or therapeutic radiation therapy
* currently enrolled in or has not yet completed at least 30 days since ending other investigational device or therapy, or subject is receiving other investigational agent(s)
* active infection requiring treatment within 1 week before enrollment
* undergone major surgery within 4 weeks before enrollment or recovering from prior surgery
* past or current history of another neoplasm, except for curatively treated non-melanoma skin cancer, carcinoma in situ of the cervix and other primary solid cancer with no known active disease present and no curative treatment administered for the last 3 years
* known allergy or sensitivity to any of the excipients in the investigational product to be administered
* pregnant or is breast feeding
* not consenting to use adequate contraceptive precautions during the course of the study and for 6 months after the last administration of investigational product:

  * female subjects who are not post-menopausal (no menstrual period for a minimum of 12 months at study entry) or documented surgically sterile will not be bound to this exclusion
* previously treated with AMG 102
* previously enrolled into this study
* will not be available for follow-up assessments
* has other disorders that compromises the ability of the subject to give written informed consent and/or comply with study procedures
* unable to begin protocol specified treatment within 3 days after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the objective response rate in subjects with advanced renal cell carcinoma receiving AMG 102 treatment | 9 weeks from first dose of AMG 102

SECONDARY OUTCOMES:
To estimate the overall survival and progression free survival rates in this population | 8 week intervals
To assess the duration of response and time to response in this population | treatment period
To assess the pharmacokinetics of AMG 102 in subjects with advanced renal cell carcinoma | Weeks 1, 5, and 9
To assess the safety profile of AMG 102 in subjects with advanced renal cell carcinoma | entire study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Schoffski P, Garcia JA, Stadler WM, Gil T, Jonasch E, Tagawa ST, Smitt M, Yang X, Oliner KS, Anderson A, Zhu M, Kabbinavar F. A phase II study of the efficacy and safety of AMG 102 in patients with metastatic renal cell carcinoma. BJU Int. 2011 Sep;108(5):679-86. doi: 10.1111/j.1464-410X.2010.09947.x. Epub 2010 Dec 13. PMID 21156020
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com